CLINICAL TRIAL: NCT01628484
Title: Comparison of the Influence of Different Skin Conditions on the Allergic Skin Reactivity to Epicutaneous Allergen Exposure
Brief Title: Physiological Study to Determine the Allergic Skin Activity After Different Skin Preparation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SkinPrep
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Birch Pollen Allergy
MeSH Terms: interventions — PittCoVacc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skin Preparation Testing (Other): The methodology of this study is an intra-individual comparison. Each study participant is treated with three skin preparation techniques (pricking, tape stripping, microneedle array)on both volar forearms.
  Interventions: Other: prick lancet; Other: Tape stripping; Other: Microneedle

INTERVENTIONS:
Other: prick lancet — For the pricking skin preparation, sterile prick lancets for 1mm point skin testing will be used. They are used for allergy diagnostics in daily routine.
  Other Names: Prick Lancet; Worcestershire, UK; distr. by Stallergenes®.
Other: Tape stripping — For the tape stripping in the skin preparation test conventional self adhesive tape by Tesafilm® is used.
  Other Names: Tesafilm
Other: Microneedle — To induce a large number of microchannels with a maximal depth of 150µm into the cornea layer a small patch of 351 tiny needles is used, which is on the market in the US and is intended for preparing the skin for transdermal application of topical dermatology products.
  Other Names: solid Microstructured Transdermal System (sMTS) by 3M®

SUMMARY:
The objectives of this monocentric investigator initiated exploratory clinical trial is to optimize allergen delivery across the epidermal barrier. The cornified outer epidermal layers represent the main barrier towards entry into the viable epidermal layers. In the latter we aim to target the allergen for uptake by professional antigen presenting cells, called Langerhans cells. At the same time as little allergen as possible should be delivered to the dermis. The latter contains a high density of sensitized mast cells eliciting local reactions and also a high density of blood vessels which could lead to systemic distribution of allergen and therefore to systemic allergic reactions.

In birch pollen allergic individuals we will compare different methods of preparing the skin before application of the allergen. We will subsequently apply titrated allergen doses to the prepared skin areas to determine at which dose we start observing mast cell degranulation manifesting as hives.

This will allow for determination of the maximal tolerated allergen dose for each skin preparation method.

The skin preparation methods compared will be:

* Single pricking with prick lancet (Entaco LTD., Redditch, Worcestershire, UK, distributed by Stallergenes®).
* Tape stripping with conventional adhesive Tape (Tesa-film®).
* Microchanneling with Micro Needle Patch (Micro Skin System, 3M®). The methods are strongly connected to routine diagnostics of allergies with low risk associated.

The clinical trial protocol has been submitted to the local Ethics Committee.

This comparison of skin preparation methods and the determination of the maximal tolerated allergen dose will help us to further improve epicutaneous allergen immunotherapy, which has the potential to make allergen specific immunotherapy not only considerably shorter and safer, but also more convenient for patients. Skin preparation by microneedle patches is significantly less painful than conventional injection and can be self administered. This should help improve the acceptance of allergen specific immunotherapy, as well as treatment compliance.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION The prevalence of allergic diseases has been continuously increasing, reaching a prevalence of up to 30% in industrialized countries. In Switzerland, about 2 million people are affected by IgE-mediated allergies as reported by the Swiss Center for Allergy, Skin and Asthma and the Swiss Society for Allergology and Immunology (SSAI). By subcutaneous injections of gradually increasing allergen doses, conventional subcutaneous SIT (SCIT) is found to reduce the inappropriate T-helper (Th) 2 responses and IgE production. Due to the risk of systemic allergic side effects, the typical therapy duration of 3-5 years and the requirement of 50-80 injections, patient acceptance of SCIT is low and less than 5% of allergy patients choose to undergo SCIT. A recently rediscovered route of allergen administration is via the epidermis in a procedure called epicutaneous immunotherapy (EPIT).

The skin is an attractive administration route for immunotherapy being both easily accessible as well as playing an important role in the immune system consisting of keratinocytes, Langerhans cells (LC), dermal dendritic cells (DC). A major challenge in EPIT is to overcome the physiological barrier function of the skin. In order to deliver the allergen to the immunological effector cells in the skin, the allergen must be transported through the outermost keratinized layer of the epidermis, called the stratum corneum. The stratum corneum is 10-20μm thick and impermeable for molecules greater than 500 Da. Proteins, such as allergens, do not passively permeate across the skin and therefore enhancement strategies are needed to enable this transfer. Advances in microtechnology might contribute to improve the situation by allowing for the miniaturization of mechanics and structures. As the stratum corneum is only 10-20μm thick, it has been proposed by Henry et al., that microneedles as small as a few tens to a few hundreds of microns, could be used to penetrate the stratum corneum.

Such new methods of overcoming the skin barrier raise the question of the influence of different types of skin injury patterns on the allergic skin reactivity. Namely, how important is the role of the exposed area (microneedles), the depth of injury (skin pricking) and the keratinocyte activation. This physiological question is in the focus of this study.

PRODUCTS In order to investigate the physiological reactions concerning different skin conditions and allergen exposition the following products/techniques have been chosen for the purpose of inducing different skin conditions in a reproducible way.

Prick lancet:

For the pricking skin preparation, sterile prick lancets for 1mm point skin testing will be used: prick lancet, produced by Entaco LTD., Redditch, Worcestershire, UK and distributed by Stallergenes®. They are used for allergy diagnostics in daily routine.

Adhesive tape:

For the tape stripping skin preparation a conventional tape will be used (Tesafilm®).

Microneedle array:

To induce a large number of microchannels with a maximal depth of 150μm into the cornea layer,the solid Microstructured Transdermal System (sMTS) by 3M® will be used. This system is a small patch of 351 tiny needles, which is on the market in the US and is intended for preparing the skin for transdermal application of topical dermatology products.

Epicutaneous allergen solution:

For the epicutaneous administration four ten-fold serial dilutions (10 HEP, 1 HEP, 0.1 HEP and 0.01HEP/ml) of registered allergen extracts of birch pollen (Betula verrucosa) (Soluprick®, ALK-Abelló A/S, Hørsholm, Denmark) will be used as in everyday allergy diagnostic practice. Histamine as positive control will be used at 10 mg/ml and a solution containing only the excipients will serve as negative control.

This is an open-label physiological investigation of the allergic skin reactivity to epicutaneous allergen exposition in allergic patients comparing different methods of skin preparation. The focus of the study is on the skin preparation and not on the specific allergen or allergy, but for reasons of homogeneity a single allergic disease, birch pollen allergy was chosen as the basis for the testing. In order to evaluate the effects of the different skin preparation techniques an intra-individual comparison of the skin reactivity in terms of the immediate phase I reaction to serial dilutions of birch pollen extracts was chosen. The serial dilution approach allows a dose dependent effect evaluation and determination of the mean allergen concentration yielding similar skin reactions - thus differences will be explained mainly by the different skin preparation allowing a quantitative comparison of these techniques.

HYPOTHESIS We will determine which of the three different skin preparation techniques uses higher protein concentration of allergen preparation (Ch10) eliciting a wheal area of the same size as histamine 10 mg/ml will be calculated.

The Null hypothesis therefore would be:

Ch10 is not significantly different between the three skin preparation techniques.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* 18-65 years old (male and female)
* A positive clinical history for inhalant allergy presumably due to birch pollen
* Positive screening prick test (mean wheal diameter = 3mm) to birch pollen allergen solution
* A mean wheal size of = 7mm2 obtained in the screening prick test with histamine dihydrochloride (10mg/ml)

Exclusion criteria:

* Impaired in understanding the nature, meaning and scope of the study or incapable of giving written informed consent
* Participation in another clinical trial within the last 30 days and during the present study
* Pregnancy or nursing
* Positive skin reaction in the screening prick test to NaCl
* Currently suffering from allergy symptoms
* History of systemic reactions to allergens
* Severe diseases influencing the results of the present study by discretion of the investigator
* Immunotherapy with the allergen preparation during the past two years
* Skin lesions and excessive hair-growth in the skin test areas
* Treatment with prohibited concomitant medications, with the exception of medications with local effects which will not influence the results of the skin prick tests
* Alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Wheal size of the immediate reaction in mm2. | 15 minutes

SECONDARY OUTCOMES:
Late phase response. | 3 days
  Evaluation of late phase reaction (eczema development).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kuendig, MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Zurich, Division of Dermatology, Zurich, Canton of Zurich, Switzerland